CLINICAL TRIAL: NCT03234595
Title: Everfront Biotech Co., Ltd.
Brief Title: A Phase I/IIa Study of Cerebraca Wafer Plus Adjuvant Temozolomide (TMZ) in Patients With Recurrent High Grade Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Everfront Biotech Co., Ltd. (Industry)
Collaborators: DOIT, Ministry of Economic Affairs, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFBPOLZ20141120
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Recurrent GBM
Keywords: Cerebraca Wafer; Recurrent high-grade glioma; Astrocytoma; Glioblastoma; IDH wild type; MGMT unmethylation (chemoresistance)
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): There is 1 treatment arm with 4 dose cohorts in Phase I and 1 treatment arm in Phase IIa.
  Interventions: Drug: Cerebraca wafer

INTERVENTIONS:
Drug: Cerebraca wafer — Eligible patients will receive Cerebraca wafer implantation with adjuvant temozolomide (TMZ) for the safety and efficacy in this study. At Phase I, the MTD will be determined by DLT. At Phase IIa, up to 12 evaluable patients will be enrolled for the efficacy and safety of Cerebraca wafer implantation. At Phase IIa, the cavity surface after tumor removal will be maximally covered by Cerebraca wafer without exceeding the MTD defined at Phase I. Patients in Phase I receive treatment as designed for Phase IIa, the data will be incorporated into Phase IIa to reduce the patient number. The overall patient number in this study is therefore between 2 to 36 evaluable patients.

SUMMARY:
Cerebraca Wafer (75 mg [(Z)-n-butylidenephthalide]) is designed for surgical combination to treat glioblastoma (GBM) diseases. High-grade glioma includes GBM (Grade IV, isocitrate dehydrogenase 1 [IDH1] wild-type) and anaplastic astrocytoma (Grade IV and Grade III, IDH1 mutation). Among these, GBM is the most common and aggressive brain tumor. Patient suffering from GBM usually develops symptoms such as headaches, seizures, memory loss, and changes in behavior in its early phase. At later stages, patients may encounter loss of movement and sensation, language dysfunction, and cognitive impairments depending on location and size of the tumor. The average survival of recurrent GBM patients is 6 to 9 months regardless of the use of current available therapies.

The clinical trial aimed to evaluate the safety and efficacy profiles of Cerebraca Wafer plus adjuvant TMZ in patients with recurrent GBM. Additionally, the study sought to determine the maximum tolerated dose (MTD) of Cerebraca Wafers. This study specifically examined the safety of the intended dose of 6 wafers.

DETAILED DESCRIPTION:
* This is a first-in-human, open-label, one-arm, Phase I/IIa study to investigate the safety and efficacy of Cerebraca Wafer with adjuvant TMZ treatment in patients with recurrent high-grade glioma. Eligible participants are to receive Cerebraca Wafer implantation as well as TMZ treatment.
* Phase I is a typical dose escalation study utilizing traditional 3+3 study design. There are 4 dose levels in this stage. DLT is to be assessed during the Phase I to evaluate the safety and tolerance of Cerebraca Wafer and to determine the MTD. Data and Safety Monitoring Board (DSMB) meetings are held before dose escalation and for MTD determination.
* In Phase IIa, participants are to be enrolled for assessment of the efficacy and safety. The cavity surface after tumor removal is maximally covered by Cerebraca Wafer without exceeding the MTD defined in Phase I. Data collected from participants in Phase I receiving treatment as designed for Phase IIa are incorporated into Phase IIa to reduce the participant number. The study consists of 2 periods:

  1. Main Study Period (including Screening Visit [up to 30 days] and Contiguous and Intermitting Visits [overall 24 weeks])
  2. Extended Period (including Follow-up Visits [every 8 weeks])

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, age ≥ 20 years old
2. Patient has diagnosed recurrent high grade glioma, including anaplastic astrocytoma and glioblastoma multiforme
3. Patients have enough cavity after glioma resection for planned number of wafer implantation (by Investigator's judgment)
4. Patients have unilateral single focus of tumor in cerebrum
5. Patients have the 1st time recurrence of glioma
6. Patients undergone standard therapy for their prior glioma episode; for patients with anaplastic astrocytoma, the prior standard therapy should include surgical resection, radiation and adjuvant temozolomide (or PCV [procarzine, lomustine and vincristine]; for patients with glioblastoma multiforme the prior standard therapy should include surgical resection, radiation and adjuvant temozolomide
7. Patients with Karnofsky Performance Score (KPS) ≥ 50
8. Patients are recovered from toxicities from prior systemic therapies and have adequate hematopoietic function at screening and before using study medication

   * Absolute neutrophil count (ANC) ≥ 1,000 cells /mm3
   * Platelets ≥ 100,000 /mm3
   * Total white blood cell (WBC) ≥ 2,500 cells /mm3
   * Total bilirubin ≤ 2.5 mg/dL
   * AST ≤ 4 x ULN
   * ALT ≤ 4 x ULN
   * ALP ≤ 5 x ULN
   * Creatinine ≤ 2.0 mg/dL
   * GFR ≥ 30 ml/min/1.73m2
9. Patient with no or mild organ impairment
10. Patients who are eligible and able to participate in the study and accept to enter the study by signing written informed consent forms
11. Patients agrees not to use food supplementary or dietary that contains Angelica sinensis after Screening Visit to Day 21
12. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use appropriate contraception method(s) for at least 4 weeks after Cerebraca wafer treatment and TMZ treatment (whichever is longer) shown below.

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Combination of any two of the following (a+b or a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Phase IIa The inclusion criteria for Phase IIa is the same as in Phase I

Exclusion Criteria:

Phase I and IIa

1. Patient who has participated in other investigational studies within 4 weeks prior to receive Cerebraca wafer
2. Patient with known or suspected hypersensitivity to Cerebraca wafer, TMZ or the excipient
3. Patient has tumor that cannot be surgically removed without significantly affecting vital function
4. Patient's glioma locates in the area that is not suitable for Cerebraca wafer implantation
5. Patient has external-beam radiation therapy within 4 weeks before study entry
6. Patient has other severe and/or life-threatening disease(s) with life expectancy less than 12 months
7. Patient has immuno-compromised condition, or is with known autoimmune conditions or is human immunodeficiency virus (HIV) seropositive.
8. Patient with medical, social or psychological factors interfering with compliance of the study
9. Patient has on-going moderate to severe organ impairment other than study indication that may confound the efficacy evaluation, safety evaluation or usage of TMZ
10. At Phase I, patient is planning to use strong cytochrome P450 modulator.
11. Female patients are lactating, pregnant, or planned to be pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of Cerebraca Wafer by dose limiting toxicity (DLT) in patients with recurrent high-grade glioma. | 2 year
  MTD and DLT
To evaluate the efficacy profiles of Cerebraca Wafer in patients with recurrent high-grade glioma. | 2 year
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Hualien Tzu Chi Hospital, Hualien City
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei